CLINICAL TRIAL: NCT03710915
Title: A Phase I Study of Single-centre, Open-label Clinical Trial to Evaluate HG146 Capsule in the Treatment of Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of HG146 Capsule in Chinese Subjects with Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: HitGen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HG146-I-CRP-1.0
Record Dates: First submitted 2018-09-29; First posted 2018-10-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma; Relapsed and Refractory Multiple Myeloma
Keywords: HDAC inhibitor; Dose escalation; HG146
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Intervention Model Description: Drug: HG146 capsule HG146 capsule is a histone deacetylase inhibitor (HDAC inhibitor) for the treatment of multiple myeloma.
  Other Name: HG280146, HG0146, HG280146, HG280146-P1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG146 capsule treat multiple myeloma (Experimental): Experimental: 5/10/15/20 mg HG146 capsule 5 mg starting dose taken orally on Day 1, 3, 5, 7, 9, 11, 13 of each cycle, and off drug for 8 days (3 weeks).
  Intervention: Drug: HG146 capsule
  Interventions: Drug: HG146

INTERVENTIONS:
Drug: HG146 — HG146 will be administered every other day for 14 days, followed by 1 week off the drug with each treatment cycle of 21-days.
  Other Names: HG280146, HG0146, HG280146, HG280146-P1

SUMMARY:
This study is designed to evaluate the tolerability and safety of HG146 capsule in patients with multiple myeloma.

DETAILED DESCRIPTION:
This study is mainly designed to evaluate the tolerability and safety of HG146 capsule in patients with multiple myeloma. Secondly, to get pharmacokinetic data and preliminary efficacy of HG146 capsule in human.

This study adopts the traditional design of "3 + 3" dose escalation. The starting dose is 5 mg and subsequent dose group is respectively for 10, 15 and 20 mg. For each dosing group, subjects are administered orally HG146 every other day for two weeks, followed by one week of rest with 21-day as one treatment cycle. Patients will be treated for 4 cycles or disease progression or unacceptable toxicities, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma requiring systemic therapy (International Myeloma Working Group [IMWG]) and 2 cycles of treatment including proteasome inhibitors and/or immunomodulators.
* Serum M protein≥ 10.0g / L, or urine M protein ≥ 200mg / 24h.
* Not suitable for autologous bone marrow transplantation or refuse autologous bone marrow transplantation or relapse after autologous bone marrow transplantation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or 2.
* Expected survival of ≥3 months.
* Hemoglobin ≥ 80 g/L, Platelet≥75×10^9/L, Absolute Neutrophil Count≧1.0×109/L (1000 cells/mm3), Prothrombin time(PT) and activated partial thromboplastin time ≤ 2 x Upper Limit of Normal (ULN).
* Bilirubin in serum<1.5*ULN (2.0mg/dL/20mg/L/34.2μmol/L); glutamic-pyruvic transaminase (ALT) and/or Aspartate Aminotransferase (AST)≤3*ULN (upper limit of normal).
* Normal electrocardiogram, echocardiography and myocardial enzyme spectrumCalibration of blood calcium concentration≤ULN.
* Men and women, Non-pregnant women who did not consider giving birth during the trial or five years after the end of the trial.
* The patient is able to swallow the capsule.
* Patients must provide written consent.

Exclusion Criteria:

* Severe allergies to the study drug or any of its excipients.
* The possibility of gene toxicity, mutagenesis and teratogenicity.
* Men and women who did not have sperm or egg cells stored in vitro before the trial and who planned to have children again within five years.
* Pregnant or lactating women.
* Perform autologous bone marrow transplantation 3 months before admission.
* Receive allogeneic bone marrow transplantation.
* Use HDAC inhibitors before.
* Two weeks prior to admission, received radiotherapy or bone marrow suppressive chemotherapy or biological treatment.
* Patients with history of other malignant tumors, except the tumor is in remission and has not been treated for at least 5 years.
* Patients with dysphagia or oral absorption disorder.
* The investigators determine the conditions not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of HG146 | Up to 3 months
  To determine the maximum tolerated dose of HG146 in relapsed and refractory multiple myeloma patients.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | In cycle 1 (each cycle is 21 days)
  To determine the Peak Plasma Concentration of HG146.
Area under the plasma concentration versus time curve (AUC) | In the middle of cycle 1 (each cycle is 21 days)
  To determine the Area under the plasma concentration versus time curve of HG146.
Time of Peak Concentration (Tmax) | In the middle of cycle 1 (each cycle is 21 days)
  To determine the time of peak concentration of HG146.
Half life (T1/2) | In the middle of cycle 1 (each cycle is 21 days)
  To determine the half-life of HG146.
Incidence of adverse events related to treatments | Up to 21 days after last dose
  To evaluate the incidence of adverse events that are related to treatments in relapsed and refractory myeloma patients.
Incidence of laboratory abnormalities related to treatments | Up to 1 month after last dose
  To evaluate the incidence of laboratory abnormalities that are related to treatments in relapsed and refractory myeloma patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Liu, M.D., Principal Investigator — The West China Hospital of Sichuan University
Locations (1):
- HitGen Inc, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang B, Lu J, Wang X, Xiao Y, Zhao Y, Huang H, Liu J, Chen M, Gu J, Yuan S, Zheng D, Li Y, Huang X, Li J. Prognostic value of lactate dehydrogenase in Chinese patients with newly diagnosed transplant eligible multiple myeloma. Leuk Lymphoma. 2017 Jul;58(7):1740-1742. doi: 10.1080/10428194.2016.1252975. Epub 2016 Nov 23. No abstract available. PMID 27881052
- [Background] Lu J, Lu J, Chen W, Huo Y, Huang X, Hou J; Chinese Medical Doctor Association Hematology Branch. Clinical features and treatment outcome in newly diagnosed Chinese patients with multiple myeloma: results of a multicenter analysis. Blood Cancer J. 2014 Aug 15;4(8):e239. doi: 10.1038/bcj.2014.55. PMID 25127393
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Durie BG, Salmon SE. A clinical staging system for multiple myeloma. Correlation of measured myeloma cell mass with presenting clinical features, response to treatment, and survival. Cancer. 1975 Sep;36(3):842-54. doi: 10.1002/1097-0142(197509)36:33.0.co;2-u. PMID 1182674
- [Background] Palumbo A, Avet-Loiseau H, Oliva S, Lokhorst HM, Goldschmidt H, Rosinol L, Richardson P, Caltagirone S, Lahuerta JJ, Facon T, Bringhen S, Gay F, Attal M, Passera R, Spencer A, Offidani M, Kumar S, Musto P, Lonial S, Petrucci MT, Orlowski RZ, Zamagni E, Morgan G, Dimopoulos MA, Durie BG, Anderson KC, Sonneveld P, San Miguel J, Cavo M, Rajkumar SV, Moreau P. Revised International Staging System for Multiple Myeloma: A Report From International Myeloma Working Group. J Clin Oncol. 2015 Sep 10;33(26):2863-9. doi: 10.1200/JCO.2015.61.2267. Epub 2015 Aug 3. PMID 26240224
- [Background] Lu J, Lee JH, Huang SY, Qiu L, Lee JJ, Liu T, Yoon SS, Kim K, Shen ZX, Eom HS, Chen WM, Min CK, Kim HJ, Lee JO, Kwak JY, Yiu W, Chen G, Ervin-Haynes A, Hulin C, Facon T. Continuous treatment with lenalidomide and low-dose dexamethasone in transplant-ineligible patients with newly diagnosed multiple myeloma in Asia: subanalysis of the FIRST trial. Br J Haematol. 2017 Mar;176(5):743-749. doi: 10.1111/bjh.14465. Epub 2017 Jan 20. PMID 28106903